CLINICAL TRIAL: NCT06921057
Title: Effects of Exergames on Muscle Strength and Lung Function in Elderly
Brief Title: Effects of Exergames on Muscle and Lung Function in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Chen Yen-Huey, associate professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202301151B0
Record Dates: First submitted 2025-03-31; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Aging
MeSH Terms: interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exergame (Experimental): playing exergame 30 min/session, 2 sessions/ week, for 8 weeks.
  Interventions: Other: exergame
- Control (No Intervention): remain regular activities for 8 weeks.

INTERVENTIONS:
Other: exergame — playing exergames
  Arms: exergame

SUMMARY:
The goal of this study is to examine the effects of 8-weeks exergames program on pulmonary function, muscle strength and cognitive function in elderly.

Participants will:

Play exergame 30min/session, 2 sessions/week or remained regular daily activities for 8 weeks.

DETAILED DESCRIPTION:
Subjects who are older than 60 years will be assigned to exergame group or control group randomly.

Exergame group: Subjects will receive exergame program 30min/session, 2 sessions/week for 8 weeks.

Control group: Subjects remain regular daily activities for 8 weeks. Both groups receive pre- and post- measurements. The measurements included assessment of muscle strength and lung function.

ELIGIBILITY:
Inclusion Criteria:

1. age > 60 years,
2. sufficient cognitive capacity to provide informed consent,
3. ability to understand and speak Chinese or Taiwanese.

Exclusion Criteria:

1. medical conditions prohibiting physical exercise
2. physical or cognitive disabilities preventing participation in or comprehension of the exergame.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
forced expiratory volume at 1 sec (L) | week 0 and week 8
  forced expiratory volume at 1sec
forced expiratory volume at 1 sec (%) | week 0 and week 8
  percentage of forced expiratory volume at 1sec predicted value
forced vital capacity(L) | week 0 and week 8
  forced vital capacity
forced vital capacity(%) | week 0 and week 8
  percentage of forced vital capacity predicted value
arm curl test | week 0 and week 8
  measurement upper arm muscle strength
hand grip strength | week 0 and week 8
  measurement upper arm muscle strength
Mini-Mental State Examination | week 0 and week 8
  assessment of cognitive function
Montreal Cognitive Assessment | week 0 and week 8
  assessment of cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Huey Chen, PhD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: 2025/01-2025/06
Access Criteria: Data are available from the PI upon reasonable request.